CLINICAL TRIAL: NCT07023484
Title: Personalized Timing of Interval Debulking Surgery Based on KELIM After Neoadjuvant Chemotherapy in Advanced Ovarian Cancer - a Multicenter Randomized Phase II Non-inferiority Trial (PRESELECT-I Trial)
Brief Title: Personalized Timing of Interval Debulking Surgery in Advanced Ovarian Cancer
Acronym: Preselect-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); United Christian Hospital (Other); Pamela Youde Nethersole Eastern Hospital (Other); The University of Hong Kong-Shenzhen Hospital (Other); Sun Yat-sen University Cancer Centre (Unknown)
Responsible Party: Principal Investigator, Dr. Ka-Yu Tse, Prof., The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 24-746; HKUCTR-3092 (Registry Identifier: HKU Clinical Trials Registry)
Record Dates: First submitted 2025-06-07; First posted 2025-06-17 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: advanced; ovarian cancer; fallopian tube cancer; primary peritoneal cancer; neoadjuvant chemotherapy; interval debulking surgery; kelim
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: non-inferiority randomised trial
Who Masked: Outcomes Assessor
Masking Description: Completeness of resection is assessed by independent surgeon
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard clinical practice (Active Comparator): Participants will follow the standard practice and receive 3-6 cycles of neoadjuvant chemotherapy, followed by radiological assessment and interval debulking surgery.
  Interventions: Drug: Carboplatin plus Paclitaxel; Procedure: Interval debulking surgery
- Personalised management (Experimental): Patients will be managed based on CA-125 ELIMination Rate Constant K (KELIM) at the neoadjuvant setting.
  Interventions: Diagnostic Test: KELIM; Drug: Carboplatin plus Paclitaxel; Procedure: Interval debulking surgery

INTERVENTIONS:
Diagnostic Test: KELIM — (i) Patients with KELIM =>1 will receive radiological assessment and undergo internal debulking surgery if the disease is operable. (ii) Patients with KELIM <1 will have alternative management, such as addition of bevacizumab or changing to dose-dense chemotherapy, and defer the interval debulking surgery
  Arms: Personalised management
Drug: Carboplatin plus Paclitaxel — Neoadjuvant chemotherapy
Procedure: Interval debulking surgery — Interval debulking surgery

SUMMARY:
About 70% of epithelial ovarian cancer patients are diagnosed at advanced stage. When primary optimal surgery is not possible, neoadjuvant chemotherapy will followed by interval debulking surgery is one treatment option. However, there is no consensus on the optimal timing of the surgery. CA125 is a well-known tumor marker in ovarian cancer. Its kinetic change has been proven to correlate with the patients' response to chemotherapy and chance of optimal resection. This study aims to utilize the kinetic change of CA125 to customize the timing of surgery for individual patients and compare this with the standard clinical practice.

DETAILED DESCRIPTION:
Recruited patients will be randomised into two groups. The control group will receive treatment according to the standard clinical practice. The investigation group will have an additional CA125 at the 5th week after the first cycle of chemotherapy. CA-125 ELIMination Rate Constant K (KELIM) will be determined using online tool. Patients with KELIM =>1 will receive radiological assessment and undergo internal debulking surgery if the disease is operable. Patients with KELIM <1 will have alternative management, such as addition of bevacizumab or changing to dose-dense chemotherapy, and defer the interval debulking surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years old or older
2. Patients with Eastern Cooperative Oncology Group score 0-1 within 28 days prior to recruitment
3. Patients who can sign the informed consent
4. Patients with stage III-IV histologically or cytologically confirmed epithelial ovarian cancer (EOC), fallopian tube or primary peritoneal cancer not amenable for PDS
5. Patients who have baseline computed tomography (CT) of thorax, abdomen and pelvis.
6. Patients who are planned for neoadjuvant chemotherapy (NACT) using 3-weekly carboplatin and paclitaxel. Those who have received one cycle of NACT may be eligible if the CA125 schedule of the study group can be matched.
7. Patients who have an evaluable CA125 level at baseline (i.e., baseline level is at least 2x upper limit of normal)
8. Patients who agree for chemotherapy and interval debulking surgery (IDS) if the disease becomes operable after NACT
9. Patients with adequate hematologic, liver and renal functions for chemotherapy
10. Patients who agree to receive adjuvant chemotherapy after IDS. The total number of NACT and adjuvant chemotherapy should be four or above, up to maximum of 9 cycles.
11. Patients who have childbearing potential should practice highly effective contraception throughout the study until at least 30 days after completion of the treatment.
12. Patients must have either germline and / or somatic BRCA test, or homologous recombination deficiency (HRD) test.

Exclusion Criteria:

1. Patients who have borderline malignancy, or non-EOC like germ cell or sex cord tumor, or metastatic diseases from other origins
2. Patients with mucinous and neuroendocrine histology
3. Patients with history of other malignancies within five years
4. Patients who are eligible for primary debulking surgery (PDS)
5. Patients who cannot undergo PDS because of parametrial and/or vaginal involvement alone
6. Patients who are not fit for PDS because of medical morbidities or refusal of operation
7. Patients who have already started NACT outside the study centers, except those who have received only one cycle within 7 days and the baseline CA125 value within 3 days of NACT (normal cut-off 35 U/ml) is available
8. Patients who participate in other interventional studies
9. Patients who are pregnant or breastfeeding
10. Patients who have contraindications to platinum-based chemotherapy
11. Patents with active tuberculosis, history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) are excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 126 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete resection (CC0) rate | up to 24 weeks from randomisation
  The likelihood of CC0 in patients who undergo IDS when KELIM reaches >=1
12-month progression-free survival (PFS) rate by RECIST criteria | up to 24 months from randomisation
  PFS is defined as the time from the date of randomization until the date of progressive disease or death (whichever comes first).

SECONDARY OUTCOMES:
Chemotherapy response score (CRS) | up to 24 weeks from randomisation
  CRS of omentum removed during interval debulking surgery CRS 1, there is no or minimal tumor response; CRS 2, there is appreciable tumor response amidst viable tumor; CRS 3, there is complete or near complete response with no residual tumor or minimal irregularly scattered tumor foci seen as individual cells, cell groups or nodules up to 2 mm
Progression-free survival (PFS) by RECIST criteria | up to 5 years from randomisation
  PFS is defined as the time from the date of randomization until the date of progressive disease or death (whichever comes first).
Overall survival (OS) | Up to 5 years from randomisation
  OS is defined as the time from the date of randomization until death due to any cause.
Incidence of adverse events | up to 1 year from randomisation
  The complication rates of surgery based on the Clavien-Dindo classification and chemotherapy based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Quality-of-life scale | up to 1 year from randomisation
  Different functional scales will be assessed by questionnaires like the EORTC questionnaires where all scales range from 0-100. The higher the score, the greater the intensity of that particular item is.

OTHER OUTCOMES:
Expression of biomarkers | up to 1 year from randomisation
  Expression levels of biomarkers before and after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yu Tse, MBBS, MMedSc, PhD, FRCOG, Principal Investigator — The University of Hong Kong
Locations (6):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen
- Hong Kong (4):
  - Pamela Youde Nethersole Eastern HospitalPamela Y, Chai Wan
  - Queen Mary Hospital, Department of Clinical Oncology, Hong Kong
  - The University of Hong Kong, Department of Obstetrics and Gynaecology, Hong Kong
  - United Christian Hospital, Kwun Tong

IPD SHARING:
Plan to Share IPD: No